CLINICAL TRIAL: NCT06203899
Title: Strong Teens and Resilient Minds: School-based Depression and Suicide Prevention in Adolescents Attending Special Schools
Brief Title: Depression and Suicide Prevention in Adolescents Attending Special Schools
Acronym: STORM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ggz Oost Brabant (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL83816.091.23
Record Dates: First submitted 2023-12-14; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-10

CONDITIONS: Depressive Symptoms
Keywords: Depression; Prevention; Adolescence; Special education
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Non-blinded cluster-randomized controlled trial with two parallel conditions (experimental and control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participating adolescents receive the preventive group training Op Volle Kracht. It is an altered program for adolescents in the special educational sector, based on the eponymous program for general education. It consists of eight meetings of 45 minutes each and one short follow-up meeting each week to offer repetition. It will take place at school during school hours. A trained psychologist of the STORM approach will facilitate the training with a trained school psychologist.
  Participants will undergo a clinical interview at baseline and at 6-month follow-up to detect clinical depression, and will fill in questionnaires at baseline, post-intervention and follow-up at 6 and 12 months after intervention. Assessments will be conducted through a 30-minute self-report questionnaire.
  All teachers will be educated on how to recognize and address depressive symptoms and suicidality in adolescents (gatekeeperstraining).
  Interventions: Behavioral: Op Volle Kracht; Behavioral: Gatekeeperstraining
- Control group (Active Comparator): Participating adolescents will undergo a clinical interview at baseline to detect clinical depression, and will fill in questionnaires at baseline, 12 weeks/'post-intervention' and follow-up at 6 and 12 months 'post-intervention'. Besides, participants will undergo a second clinical interview on depressive symptoms at 6 months follow-up.
  All teachers will be educated on how to recognize and address depressive symptoms and suicidality in adolescents (gatekeeperstraining).
  Concerning Op Volle Kracht: Adolescents are offered the training after data collection of the study has ended and when the intervention has shown to be effective.
  Interventions: Behavioral: Gatekeeperstraining

INTERVENTIONS:
Behavioral: Op Volle Kracht — This is a preventive group training based on cognitive behavioural therapy for depression.
  Arms: Intervention group
Behavioral: Gatekeeperstraining — This is a training for teachers to detect and address depressive symptoms and suicidality in their students .

SUMMARY:
Depression is a major public health concern. In Dutch adolescents, the prevalence of major depressive disorder is estimated at 3.8%, and one in five adolescents report depressive symptoms. Depression is a risk factor in adolescent suicide. School-based prevention programs, for example the STORM approach, are effective in decreasing depressive symptoms among adolescents with elevated depressive symptoms at screening. However, not all adolescents attend general education. In the Netherlands, 7% of all adolescents enters special education (voortgezet speciaal onderwijs and prakijkonderwijs). They form a vulnerable subgroup concerning developing depressive symptoms and suicidality. To adapt and implement programs for these students, is complex yet crucial. This study aims to screen adolescents, offer them a prevention program to prevent the onset or continuation of depression and evaluate the effectiveness of this program. It is a randomised controlled trial with two conditions. The main study parameter is depressive symptomatology. Secondary study parameters are suicidality, anxiety and somatic complaints.

Eligible students enter the second or third grade of special education, presenting elevated depressive symptoms. All adolescents will be screened for depressive and suicidal symptoms. Those reporting suicidality will be guided to specialised care, together with their parents. Adolescents with elevated depressive symptoms in the experimental condition will be offered the CBT-based preventive group training Op Volle Kracht in their school setting. The control condition consists of monitoring, and is offered the training if the intervention has shown to be effective. Participants will fill in longitudinal measurements. At all times, adolescents will be guided to mental health care if necessary. Furthermore, teachers in all participating schools will attend a training on how to detect and address depressive and suicidal symptoms among adolescents.

The potential value of the study is that we can offer adolescents in the special educational sector a prevention program that is proven to be effective. In order to achieve this goal we need to evaluate the effectiveness of this prevention program in this target group. We are of opinion, however, that the risks associated with participation can be considered negligible. It is specifically aimed at depressive symptoms, within a population which receives care for other problems.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents are in their second or third year of secondary education, ór adolescents will reach the age 14 or 15 in this academic year.
* Score above cut-off on depression symptom questionnaire (≥ 14 on the CDI-2; Bodden et al. (2016)).

Exclusion Criteria:

* Adolescents who score 2 on item 8 of the CDI-2 or ≥ 23 on the VOZZ-screen (Kerkhof et al., 2015).
* Clinical depression based on the clinical interview at baseline ADIS-C (Silverman & Albano, 1996).
* Absence of parental permission.
* Adolescent already receiving treatment for depressive symptomatology.
* Insufficient knowledge of the Dutch language.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 236 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms in children and adolescents | Depressive symptoms will be measured at the screening, at T0 (baseline), T1 (12 weeks), T2 (6 months), and T3 (12 months).
  Depressive symptoms in children and adolescents will be measured with the CDI-2 (Bodden et al., 2016; Kovacs, 2011). The CDI-2 contains 28 items, each consisting of three statements graded in severity from 0 to 2. This instrument has good internal consistency and convergent validity (Bae, 2012). The use of the CDI-2 for screening purposes is in accordance with the Dutch multidisciplinary guidelines for depression among youth (Richtlijnen jeugdhulp en jeugdbescherming, 2023). Suicidality will be measured with item 8 of the CDI-2. In case children score 2 on this present item, they will be seen by a health professional and eventually redirected to mental health care. Parents will be informed.

SECONDARY OUTCOMES:
The presence of a clinical depression | The presence of a clinical depression will be measured at T0 (baseline) and T2 (6 months)
  he presence of a clinical depression is measured by a clinical interview using the Anxiety Disorder Interview Schedule for Children, ADIS-C (Silverman & Albano, 1996). The study will only include the section of affective disorders. The purpose of this interview is to investigate if children meet the criteria of a depression. If participants meet the criteria of a depression, the severity will be determined using the checklist of the multidisciplinary guidance depression youth. Adolescents with a moderate - severe depression will be excluded from this study and redirected to mental health care.
Suicidality | Suicidality will be measured at the screening, at T0 (baseline), T1 (12 weeks), T2 (6 months), and T3 (12 months).
  Suicidality will be measured with the VOZZ-screen (Kerkhof et al., 2015). This questionnaire contains 10 questions regarding thoughts and actions about life, self-harm and suicide. Items are rated on a 5-point scale. Children with score 23 or above will redirected to a health professional and eventually redirected to mental health care. Parents will be informed. This procedure is equal to the procedure when children score 2 on item 8 of the CDI-2
Parent-reported depressive symptoms | Parent-reported depressive symptoms will be measured at T0 (baseline), T1 (12 weeks), T2 (6 months), and T3 (12 months).
  Parent-reported depressive symptoms are measured with the CDI-2 parent-report questionnaire consisting of 17 items. Parents indicate the presence of each symptom in the past two weeks on a 4-point-scale (Bodden et al., 2016; Kovacs, 2011).
Anxiety symptoms | Anxiety symptoms will be measured at T0 (baseline), T1 (12 weeks), T2 (6 months), and T3 (12 months).
  Anxiety symptoms are measured by using the RCADS-25 self-report questionnaire (Chorpita et al., 2000). Only items concerning anxiety will be used; the anxiety scale of the RCADS-25 show great psychometric properties (Klaufus et al., 2020). It is used in children 8 to 18 years old. Items are rated on an 4-point scale concerning prevalence.
Parent-reported anxiety symptoms | Anxiety symptoms will be measured at T0 (baseline), T1 (12 weeks), T2 (6 months), and T3 (12 months).
  Anxiety symptoms are measured by using the RCADS-25 parent questionnaire (Chorpita et al., 2000). Only items concerning anxiety will be used; the anxiety scale of the RCADS-25-P show great psychometric properties (Klaufus et al., 2020). It is used in children 8 to 18 years old. Items are rated on an 4-point scale concerning prevalence.
Somatic symptoms | Somatic symptoms will be measured at T0 (baseline), T1 (12 weeks), T2 (6 months), and T3 (12 months).
  Somatic symptoms will be measured via the Somatic Complaint List, which consists of 11 items about physical health such as 'I feel tired'. Items are rated on a 3-point scale including never, sometimes or often. It is validated for participants 8 years and older (Jellesma et al., 2007).

OTHER OUTCOMES:
Data of school-related variable: educational history | Data will be collected at T0 (baseline).
  Data of school-related variables are obtained in collaboration with the schools, including educational history, reason for attending special schools, diagnosis (if applicable), full scale IQ.
Data of school-related variable: reason for attending special schools | Data will be collected at T0 (baseline).
  Data of school-related variables are obtained in collaboration with the schools, including educational history, reason for attending special schools, diagnosis (if applicable), full scale IQ.
Data of school-related variable: diagnosis (if appliable) | Data will be collected at T0 (baseline).
  Data of school-related variables are obtained in collaboration with the schools, including educational history, reason for attending special schools, diagnosis (if applicable), full scale IQ.
Data of school-related variable: full scale IQ | Data will be collected at T0 (baseline).
  Data of school-related variables are obtained in collaboration with the schools, including educational history, reason for attending special schools, diagnosis (if applicable), full scale IQ.
Demographic information | Data will be collected at T0 (baseline).
  Data is gathered through questionnaires.
Previous or present receipt of professional help for psychological problems. | Data will be collected at T0 (baseline) and at T3 (12 months).
  Data is gathered through questionnaires. Course adherence will be measured in terms of session attendance.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy CH Rongen, MSc, Principal Investigator — Ggz Oost Brabant
Locations (1):
- GGZ Oost Brabant, Boekel, Noordoost Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After the PhD trajectory has ended (january 2027). For the time frame of 15 years after data collection.
Access Criteria: Data may be used to replicate the study and in meta analyses. Requests will be reviewed by the principal investigator and/or the head of the research department of GGZ Oost Brabant.

REFERENCES:
- [Background] Bodden, D., Braet, C., & Stikkelbroek, Y. (2016). Children's depression inventory-2. In: hogrefe.
- [Background] Bae, Y. (2012). Test review: children's depression inventory 2 (CDI 2). In: Sage Publications: Los Angeles, CA.
- [Background] Chorpita BF, Yim L, Moffitt C, Umemoto LA, Francis SE. Assessment of symptoms of DSM-IV anxiety and depression in children: a revised child anxiety and depression scale. Behav Res Ther. 2000 Aug;38(8):835-55. doi: 10.1016/s0005-7967(99)00130-8. PMID 10937431
- [Background] Jellesma FC, Rieffe C, Terwogt MM. The Somatic Complaint List: validation of a self-report questionnaire assessing somatic complaints in children. J Psychosom Res. 2007 Oct;63(4):399-401. doi: 10.1016/j.jpsychores.2007.01.017. PMID 17905048
- [Background] Kerkhof, A., Huisman, A., Vos, C., & Smits, N. (2015). Handleiding VOZZ & VOZZ screen: Vragenlijst over Zelfdoding. Amsterdam: Vrije Universiteit Amsterdam.
- [Background] Klaufus L, Verlinden E, van der Wal M, Kosters M, Cuijpers P, Chinapaw M. Psychometric evaluation of two short versions of the Revised Child Anxiety and Depression Scale. BMC Psychiatry. 2020 Feb 5;20(1):47. doi: 10.1186/s12888-020-2444-5. PMID 32024481
- [Background] Kovacs, M. (2011). Children's Depression Inventory 2nd edition (CDI 2): Technical manual. Multi-Health Systems.
- [Background] Richtlijnen jeugdhulp en jeugdbescherming. (2023). Richtlijn stemmingsproblemen.
- [Background] Lyneham HJ, Abbott MJ, Rapee RM. Interrater reliability of the Anxiety Disorders Interview Schedule for DSM-IV: child and parent version. J Am Acad Child Adolesc Psychiatry. 2007 Jun;46(6):731-736. doi: 10.1097/chi.0b013e3180465a09. PMID 17513985
- [Derived] Rongen WCH, Creemers DHM, Spijker J, Vermulst AA, Rasing SPA. Evaluation of a school-based depression prevention approach among adolescents with elevated depressive symptoms attending special education: study protocol of a cluster randomized controlled trial. BMC Psychiatry. 2025 May 22;25(1):517. doi: 10.1186/s12888-025-06955-5. PMID 40399869